CLINICAL TRIAL: NCT02255422
Title: A Phase 2 Study of the Safety, Efficacy, and Pharmacodynamics of RTA 408 in the Treatment of Mitochondrial Myopathy (MOTOR)
Brief Title: RTA 408 Capsules in Patients With Mitochondrial Myopathy - MOTOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: RTA 408-C-1403
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: MItochondrial Myopathies
Keywords: omaveloxolone; RTA 408 capsules; mitochondrial myopathies
MeSH Terms: conditions — Mitochondrial Myopathies | interventions — omaveloxolone; ORF 50 transactivator

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- omaveloxolone Capsules 2.5 mg and 5 mg (Experimental): omaveloxolone (RTA 408) Capsules, 2.5 mg taken orally once daily for 2 weeks, then 5 mg taken orally once daily for 10 weeks
  Interventions: Drug: Omaveloxolone capsules, 2.5 mg; Drug: omaveloxolone capsules, 5 mg
- omaveloxolone Capsules 10 mg (Experimental): omaveloxolone (RTA 408) capsules, 10 mg taken orally once daily for 12 weeks
  Interventions: Drug: omaveloxolone capsules, 10 mg
- Placebo Capsules (Placebo Comparator): Placebo capsules taken orally once daily for 12 weeks
  Interventions: Drug: Placebo capsules
- omaveloxolone Capsules 20 mg (Experimental): omaveloxolone (RTA 408) Capsules, 20 mg taken orally once daily for 12 weeks.
  Interventions: Drug: omaveloxolone capsules, 20 mg
- omaveloxolone Capsules 40 mg (Experimental): omaveloxolone (RTA 408) Capsules, 40 mg taken orally once daily for 12 weeks.
  Interventions: Drug: omaveloxolone capsules, 40 mg
- omaveloxolone Capsules 80 mg (Experimental): omaveloxolone (RTA 408) Capsules, 80 mg taken orally once daily for 12 weeks.
  Interventions: Drug: omaveloxolone capsules, 80 mg
- omaveloxolone Capsules 160 mg (Experimental): omaveloxolone (RTA 408) Capsules, 160 mg taken orally once daily for 12 weeks.
  Interventions: Drug: omaveloxolone capsules, 160 mg

INTERVENTIONS:
Drug: Omaveloxolone capsules, 2.5 mg
  Other Names: RTA 408 Capsules 2.5 mg
  Arms: omaveloxolone Capsules 2.5 mg and 5 mg
Drug: omaveloxolone capsules, 5 mg
  Other Names: RTA 408 capsules, 5 mg
  Arms: omaveloxolone Capsules 2.5 mg and 5 mg
Drug: omaveloxolone capsules, 10 mg
  Other Names: RTA 408, 10 mg
  Arms: omaveloxolone Capsules 10 mg
Drug: Placebo capsules
  Arms: Placebo Capsules
Drug: omaveloxolone capsules, 20 mg
  Other Names: RTA 408 capsules, 20 mg
  Arms: omaveloxolone Capsules 20 mg
Drug: omaveloxolone capsules, 40 mg
  Other Names: RTA 408 capsules, 40 mg
  Arms: omaveloxolone Capsules 40 mg
Drug: omaveloxolone capsules, 80 mg
  Other Names: RTA 408 capsules, 80 mg
  Arms: omaveloxolone Capsules 80 mg
Drug: omaveloxolone capsules, 160 mg
  Other Names: RTA 408 capsules, 160 mg
  Arms: omaveloxolone Capsules 160 mg

SUMMARY:
Mitochondrial myopathies are a multisystemic group of disorders that are characterized by a wide range of biochemical and genetic mitochondrial defects and variable modes of inheritance. Currently there are no effective treatments for this disease. Despite the heterogeneous myopathy phenotypes, a unifying feature of mitochondrial myopathies is that the pathogenic mtDNA mutations and/or nuclear mutations of the electron transport chain invariably lead to dysfunctional mitochondrial respiration. This reduction in mitochondrial respiration leads to a reduced ability to produce cellular adenosine triphosphate (ATP), often resulting in muscle weakness, exercise intolerance, and fatigue in patients with mitochondrial myopathies.

RTA 408 is a potent activator of Nrf2 and inhibitor of NF κB (nuclear factor kappa-light-chain-enhancer of activated B cells), and thus induces an antioxidant and anti-inflammatory phenotype. Several lines of evidence suggest that Nrf2 activation can increase mitochondrial respiration and biogenesis. Collectively, available data suggest that the ability of RTA 408 to activate Nrf2 and induce its target genes could potentially improve muscle function, oxidative phosphorylation, antioxidant capacity, and mitochondrial biogenesis in patients with mitochondrial myopathies.

This study will be a randomized, placebo-controlled, double-blind, dose-escalation study to evaluate the safety of omaveloxolone (RTA 408) at various doses in patients with mitochondrial myopathies.

ELIGIBILITY:
Inclusion Criteria:

1. Have mitochondrial myopathy as evidenced by the following 2 criteria (must meet both):

   1. Have a history of exercise intolerance with or without weakness and/or progressive exercise intolerance (in which modest exercise typically provokes heaviness, weakness, aching of active muscles, or tachycardia)
   2. Have a known primary mitochondrial DNA mutation or a nuclear DNA defect that is associated with reduced activity of at least 1 mitochondrially encoded respiratory chain complex
2. Be male or female and ≥18 years of age and ≤75 years of age
3. Have no changes to exercise regimen within 30 days prior to Study Day 1 and be willing to remain on the same exercise regimen during the 16-week study period
4. Have the ability to complete maximal exercise testing
5. Have a peak workload during maximal exercise testing of ≤ 1.5 W/kg
6. Be able to swallow capsules

Exclusion Criteria:

1. Have uncontrolled diabetes (HbA1c >11.0%)
2. Have B-type natriuretic peptide level >200 pg/mL
3. Have a history of clinically significant left-sided heart disease and/or clinically significant cardiac disease
4. Have known active fungal, bacterial, and/or viral infection, including human immunodeficiency virus or hepatitis virus (B or C)
5. Have known or suspected active drug or alcohol abuse
6. Have clinically significant abnormalities of clinical hematology or biochemistry, including but not limited to elevations greater than 1.5 times the upper limit of normal of aspartate aminotransferase, alanine aminotransferase, or creatinine
7. Have any abnormal laboratory test value or serious pre-existing medical condition that, in the opinion of the investigator, would put the patient at risk by study enrollment
8. Have taken any of the following drugs within 7 days prior to Study Day 1 or plan to take any of these drugs during the time of study participation:

   1. Sensitive substrates for cytochrome P450 2C8 or 3A4 (e.g., repaglinide, midazolam, sildenafil)
   2. Substrates for p-glycoprotein transporter (e.g., ambrisentan, digoxin)
9. Have participated in any other interventional clinical study within 30 days prior to Study Day 1
10. Have a cognitive impairment that may preclude ability to comply with study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - UCLA, Los Angeles, California
  - Mass General Hospital, Boston, Massachusetts
  - Akron Children's Hospital, Akron, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Insitute for Exercise & Environmental Medicine, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Medical School at Houston, Houston, Texas
- Neuromuscular Clinic, Rigshospitalet, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Madsen KL, Buch AE, Cohen BH, Falk MJ, Goldsberry A, Goldstein A, Karaa A, Koenig MK, Muraresku CC, Meyer C, O'Grady M, Scaglia F, Shieh PB, Vockley J, Zolkipli-Cunningham Z, Haller RG, Vissing J. Safety and efficacy of omaveloxolone in patients with mitochondrial myopathy: MOTOR trial. Neurology. 2020 Feb 18;94(7):e687-e698. doi: 10.1212/WNL.0000000000008861. Epub 2020 Jan 2. PMID 31896620

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 5-May-2015, last patient completed 30-Nov-2017
Groups:
- Placebo: Placebo capsules administered orally once daily for 12 weeks
- Omaveloxolone Capsules 2.5 and 5 mg: Omaveloxolone (RTA 408) 2.5 mg capsules administered orally once daily for 2 weeks then 5mg administered orally once daily for 10 weeks
- Omaveloxolone Capsules 10 mg: Omaveloxolone (RTA 408) 10 mg capsules administered orally once daily for 12 weeks
- Omaveloxolone Capsules 20 mg: Omaveloxolone (RTA 408) 20 mg capsules administered orally once daily for 12 weeks
- Omaveloxolone Capsules 40 mg: Omaveloxolone (RTA 408) 40 mg capsules administered orally once daily for 12 weeks
- Omaveloxolone Capsules 80 mg: Omaveloxolone (RTA 408) 80 mg capsules administered orally once daily for 12 weeks
- Omaveloxolone Capsules 160 mg: Omaveloxolone (RTA 408) 160 mg capsules administered orally once daily for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Omaveloxolone Capsules 2.5 and 5 mg | Omaveloxolone Capsules 10 mg | Omaveloxolone Capsules 20 mg | Omaveloxolone Capsules 40 mg | Omaveloxolone Capsules 80 mg | Omaveloxolone Capsules 160 mg
Started | 13 | 6 | 6 | 6 | 6 | 6 | 10
Completed | 13 | 6 | 5 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 53 patients were included in the baseline population
Groups:
- Omaveloxolone Capsules 2.5 and 5 mg: Omaveloxolone (RTA 408) 2.5 mg capsules administered orally once daily for 2 weeks then 5 mg administered orally once daily for 10 weeks
- Omaveloxolone Capsules 160 mg: Omaveloxolone (RTA 408) 160 mg capsules administered once daily for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | Omaveloxolone Capsules 2.5 and 5 mg | Omaveloxolone Capsules 10 mg | Omaveloxolone Capsules 20 mg | Omaveloxolone Capsules 40 mg | Omaveloxolone Capsules 80 mg | Omaveloxolone Capsules 160 mg | Total
Number analyzed (Participants) | 13 | 6 | 6 | 6 | 6 | 6 | 10 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.1 (11.86) | 52.3 (9.61) | 49.8 (14.05) | 45.5 (14.08) | 45.2 (4.71) | 30.7 (10.25) | 39.8 (15.27) | 42.9 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 3 | 4 | 5 | 4 | 6 | 32
  Male | 4 | 5 | 3 | 2 | 1 | 2 | 4 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 0 | 0 | 0 | 3 | 6
  Not Hispanic or Latino | 11 | 6 | 5 | 6 | 6 | 6 | 7 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change of Peak Workload (in Watts/kg) During Exercise Testing
Description: Cycle ergometry using a stationary recumbent bike was used to conduct maximal exercise testing. Peak work is defined as the workload at which patients reach maximal volition (defined as an inability to continue to exercise due to exhaustion). Change of peak workload during exercise testing was measured at baseline, Week 4, and Week 12. Change from baseline at Week 12 reported.
Time Frame: 12 weeks
Population: Three patients out of the 53 total were excluded from the analysis set. One each from the 20 mg arm and the 160 mg arm were excluded because they did not have post-baseline efficacy assessments. One patient from the placebo arm was excluded from analysis because their baseline maximal exercise test duration < 4 min and was not considered valid.
Measure: Least Squares Mean (Standard Error); unit: Watts/kg
Arm/Group | Placebo | Omaveloxolone Capsules 2.5 and 5 mg | Omaveloxolone Capsules 10 mg | Omaveloxolone Capsules 20 mg | Omaveloxolone Capsules 40 mg | Omaveloxolone Capsules 80 mg | Omaveloxolone Capsules 160 mg
Number analyzed (Participants) | 12 | 6 | 6 | 5 | 6 | 6 | 9
Watts/kg | 0.0090 (0.0388) | 0.020 (0.0544) | -0.0300 (0.0544) | 0.1050 (0.0596) | -0.0520 (0.0544) | -0.0660 (0.0544) | 0.0020 (0.0465)
Statistical Analysis 1: Comparison: Placebo vs Omaveloxolone Capsules 2.5 and 5 mg vs Omaveloxolone Capsules 10 mg vs Omaveloxolone Capsules 20 mg vs Omaveloxolone Capsules 40 mg vs Omaveloxolone Capsules 80 mg vs Omaveloxolone Capsules 160 mg; Primary Objective: To evaluate the change in peak work during maximal exercise testing; Test type: Superiority; p = 0.7321, Mixed Models Analysis — P-Value relates to difference in change in peak work from baseline relative to placebo for all doses pooled. Statistical significance was defined as p<0.05; Null hypothesis: wk 12 mean change from baseline ([μ RTA 408] - [μ Placebo]) in peak work = 0 w/kg. Positive change from baseline suggests improvement; LS mean difference (net) = -0.015, 95% CI 2-sided [-0.1051 to 0.0743], Standard Error of Mean 0.0446

2. Secondary Outcome: Change in 6-minute Walk Test (6MWT) Distance
Description: Patients were instructed to walk as far as they could along a marked path for 6 minutes. Distance walked was measured. If patients used a cane or walking assist device at Screening, the same walking assist device was to be used for all 6MWT assessments.
Time Frame: 6MWT was assessed at Week 4, Week 8, and Week 12 and compared to baseline
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Placebo | Omaveloxolone Capsules 2.5 and 5 mg | Omaveloxolone Capsules 10 mg | Omaveloxolone Capsules 20 mg | Omaveloxolone Capsules 40 mg | Omaveloxolone Capsules 80 mg | Omaveloxolone Capsules 160 mg
Number analyzed (Participants) | 13 | 6 | 6 | 5 | 6 | 6 | 9
Meters
  Week 4 | 40.462 (10.0539) | 19.333 (14.9658) | 18.2500 (14.9658) | -9.2000 (16.3942) | -11.6670 (14.9658) | 9.9170 (14.9658) | 10.8330 (12.2195)
  Week 8 | 24.923 (9.9381) | 12.865 (15.7374) | 33.9170 (15.1418) | 13.8000 (16.5870) | 11.0000 (15.1418) | 17.5830 (15.1418) | 28.9440 (12.3633)
  Week 12 | 29.846 (12.9276) | 17.167 (19.6519) | 17.7500 (19.6519) | 28.2000 (21.5275) | -7.833 (19.6519) | 6.2500 (19.6519) | 8.5710 (16.4721)
Statistical Analysis 1: Comparison: Placebo vs Omaveloxolone Capsules 2.5 and 5 mg vs Omaveloxolone Capsules 10 mg vs Omaveloxolone Capsules 20 mg vs Omaveloxolone Capsules 40 mg vs Omaveloxolone Capsules 80 mg vs Omaveloxolone Capsules 160 mg; Secondary Objective: To evaluate the change in 6-minute walk test (6MWT) distance at Week 4; Test type: Superiority; p = 0.0060, Mixed Models Analysis — P-value comparison is for difference in change in six minute walk distance from baseline within each dosage group relative to placebo. Statistical significance defined as p<0.05; The change from baseline in 6MWT was analyzed using the same MMRM model used for the primary efficacy endpoint. Analysis visits 0, 4, 8 and 12 used; LS mean difference (net) = -33.448, 95% CI 2-sided [-56.855 to -10.042], Standard Error of Mean 11.6473
Statistical Analysis 2: Comparison: Placebo vs Omaveloxolone Capsules 2.5 and 5 mg vs Omaveloxolone Capsules 10 mg vs Omaveloxolone Capsules 20 mg vs Omaveloxolone Capsules 40 mg vs Omaveloxolone Capsules 80 mg vs Omaveloxolone Capsules 160 mg; Secondary Objective: To evaluate the change in 6-minute walk test (6MWT) distance at Week 8; Test type: Superiority; p = 0.7325, Mixed Models Analysis — Statistical significance was defined as p<0.05. The p-value comparison is for the difference in change in 6MWD from baseline within each dosage group relative to placebo; [statistical method as in outcome 2, analysis 1]; LS mean difference (net) = -3.963, 95% CI 2-sided [-27.133 to 19.207], Standard Error of Mean 11.5300
Statistical Analysis 3: Comparison: Placebo vs Omaveloxolone Capsules 2.5 and 5 mg vs Omaveloxolone Capsules 10 mg vs Omaveloxolone Capsules 20 mg vs Omaveloxolone Capsules 40 mg vs Omaveloxolone Capsules 80 mg vs Omaveloxolone Capsules 160 mg; Secondary Objective: To evaluate the change in 6-minute walk test (6MWT) distance at Week 12; Test type: Superiority; p = 0.2210, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; [statistical method as in outcome 2, analysis 1]; LS mean difference (net) = -18.594, 95% CI 2-sided [-48.739 to 11.550], Standard Error of Mean 15.0004

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Significant adverse events are collected from the time of the first dose of study drug until the final visit or 30 days following final study dose for patients who terminated early. Both investigator assessment/questioning (systematic) and patient self reporting (non-systematic) are used in this study but were reported by the investigators as a consolidated number and are reported below as systematic.
Arm/Group | Placebo | Omaveloxolone Capsules 2.5 and 5 mg | Omaveloxolone Capsules 10 mg | Omaveloxolone Capsules 20 mg | Omaveloxolone Capsules 40 mg | Omaveloxolone Capsules 80 mg | Omaveloxolone Capsules 160 mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/6 | 1/6 | 0/6 | 1/6 | 1/6 | 1/10
Other Adverse Events (participants affected / at risk) | 11/13 | 4/6 | 6/6 | 6/6 | 6/6 | 4/6 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Omaveloxolone Capsules 2.5 and 5 mg (N=6) | Omaveloxolone Capsules 10 mg (N=6) | Omaveloxolone Capsules 20 mg (N=6) | Omaveloxolone Capsules 40 mg (N=6) | Omaveloxolone Capsules 80 mg (N=6) | Omaveloxolone Capsules 160 mg (N=10)
Tonic epileptic seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wide complex tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Right sided hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Exacerbated fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular dissociation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Omaveloxolone Capsules 2.5 and 5 mg (N=6) | Omaveloxolone Capsules 10 mg (N=6) | Omaveloxolone Capsules 20 mg (N=6) | Omaveloxolone Capsules 40 mg (N=6) | Omaveloxolone Capsules 80 mg (N=6) | Omaveloxolone Capsules 160 mg (N=10)
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 2 | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 4 | 0 | 3 | 0 | 0 | 1 | 1
Feeling abnormal (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Energy increased (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 1 | 1 | 0 | 3
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 2
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blister infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Consussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Penis injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram PR prologation (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram T wave amplitude decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Serum ferritin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Restless leg syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Head titubation (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphemia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2015-10-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT02255422/Prot_001.pdf
  • Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT02255422/SAP_000.pdf